CLINICAL TRIAL: NCT04429230
Title: A Trial of Non-invasive Brain Stimulation in Huntington's Disease
Brief Title: Non-invasive Brain Stimulation in Huntington's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115632
Record Dates: First submitted 2020-03-02; First posted 2020-06-12 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tPCS (Active Comparator): Patients of Huntington's disease will be randomly allocated into both the arms. Real tPCS arm will receive active tPCS. Then they will be crossed over to Sham tPCS arm.
  Interventions: Device: Active Transcranial pulsed current stimulation (tPCS)
- Sham tPCS (Sham Comparator): Patients of Huntington's disease will be randomly allocated into both the arms. Sham tPCS arm will receive sham tPCS. Then they will be crossed over to Real tPCS arm.
  Interventions: Device: Sham Transcranial pulsed current stimulation (tPCS)

INTERVENTIONS:
Device: Active Transcranial pulsed current stimulation (tPCS) — Active tPCS will be delivered through a pair of saline soaked (0.9% NaCl) surface sponge electrodes. Anodal stimulation will be given to brain area based on qEEG findings
  Arms: Real tPCS
Device: Sham Transcranial pulsed current stimulation (tPCS) — Electrode placement will be the same as active stimulation but the electric current will be ramped down 5 seconds after the beginning of the stimulation to make this condition indistinguishable from the experimental active stimulation.
  Arms: Sham tPCS

SUMMARY:
Huntington's disease is a disabling neurodegenerative disease. Patients present with involuntary movements of the body and cognitive symptoms like behavioral problem, difficulty in planning tasks, etc. No effective treatment is currently available for them apart from symptomatic therapy. Currently, studies are going on the effectiveness of noninvasive brain stimulation (NIBS) in neurodegenerative diseases. It is a mode of brain stimulation technique where current is delivered into the brain by placing electrodes into their scalp. Transcranial pulsed current stimulation (tPCS) is a new modality of noninvasive brain stimulation. It is a device that generates electrical impulses. The current generated from this device can stimulate underlying brain areas. The investigators have planned to study the feasibility of non-invasive brain stimulation via tPCS in these patients of Huntington's disease.

At first, the investigators will rate their involuntary body movement by a standard scale, assess arm movements by a robotic device, assess speech with standard protocol, assess brain electrophysiology by electroencephalography (EEG) and will also do gait (walking) analysis. Next, the investigators will give them 2 week (20 min/day) stimulation via real tPCS (active stimulation) or placebo (sham stimulation). After 2 weeks of stimulation, the investigators will re-assess the patient using the same tools mentioned pre-stimulation.

Each patient will receive real and placebo stimulation with a 1-month gap in between. They will not know whether they are receiving real stimulation or placebo. Assessment will be done before stimulation, after 2 week real stimulation and after 2 week sham stimulation.

DETAILED DESCRIPTION:
The investigators have planned to study the feasibility of non-invasive brain stimulation via Transcranial pulsed current stimulation (tPCS) in patients of Huntington's disease. Anodal stimulation will be given to the brain area based on quantitative electroencephalography (qEEG) findings.

Patients will be assessed clinically by standard rating scale (UHDRS) and by qEEG, KinArm and Gait - before and after 2 week (20 min per day) stimulation via tPCS or sham stimulation.

The investigators have planned to assess-

1. Speech
2. Upper limb movement via KinArm. Standard KinArm testing protocol will be used which is used universally.
3. Gait via Gait Carpet (Zeno Walkway)
4. Quantitative electroencephalography (qEEG)
5. Scale for Huntington's disease (UHDRS) tPCS will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes. Anode will be placed on the scalp over the area based on qEEG findings. Participant's speech will be recorded using a head-mounted microphone (AKGc520) and a digital recording device (Zoom H4nPro) while performing the following calibrated tasks (Calibration involves a sound level meter placed at 15cm from the mouth while talker says 'ah' at 70dBA) - a. Prolonged 'ah'. b. Rapid repetitions of the sounds "puh", "tuh", and "kuh". c. Two productions of a sentence with selected speech sounds (s, sh, p, b, t, i, a, u, ae, ai). "She saw Patty buy two poppies." d. Two times louder production of a sentence with selected speech sounds. "She saw Patty buy two poppies." e. Repetition of a continuous vowel at normal and fast rates. 'eye-eye-eyeeye- eye' without making any voice breaks or pauses". f. Read aloud a section of a standard passage - standard rainbow passage g. Monologue. Talk for two minutes about an interesting vacation (or an interesting hobby or activity). The Zeno walkway will be used in conjunction with the ProtoKinetics Movement Analysis Software (PKMAS) . The walkway contains a series of pressure sensors to detect footfalls. These data will be captured and collated via the PKMAS software, resulting in numerous spatial, temporal and pressure-related gait parameters. Timed-up-and-go (TUG) task will be used, consisting of rising from chair, walking across the 20-foot gait carpet, turning around off the carpet, walking back and sitting down. This will be performed over 3 trials. Gait analysis provides various parameters as output such as stride length, line of progression, step length, toe-offs and other temporal and spatial parameters for analysis. Neurophysiological EEG signals will be recorded, eyes-closed, no-task, using g.Nautilus g.tec wireless system. The g.tech system uses earclip reference sensors. The subject will be in a quiet place with less light or electromagnetic perturbations. During the resting state recordings, patients are seated in a comfortable arm chair and will be instructed to keep relaxed, with their eyes closed for 5 min. A paired t test will be used to compare baseline data and post tPCS data. Descriptive analysis of the neurological examination findings will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Huntington's disease diagnosed clinically or genetically proved

Exclusion Criteria:

* • Patients who can't walk even with support, like wheel chair bound patients.

  * Patients having other issues like stroke that can aggravate speech/ gait.
  * Patients who are not able to provide informed consent.
  * Patients who are unable to communicate by speech and who can't comprehend the English language.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-07 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 1 year
  Can we recruit 15 HD patients for non-invasive brain stimulation study
Feasibility of finishing the study | 1 year
  Can 15 participants finish the study
Feasibility of home based stimulation | 1 year
  Can non-invasive brain stimulation in the form of transcranial pulsed current stimulation (tPCS) be appropriately applied at home
Feasibility of network targeting | 1 year
  Can dysfunctional brain area in HD be targeted for stimulation non-invasively, using qEEG as a guide

SECONDARY OUTCOMES:
Change in UHDRS | 3 months
  The investigators will evaluate the effectiveness of tPCS in patients of Huntington's disease. The investigators will apply Unified Huntington's disease rating scale (UHDRS) pre and post stimulation. The scale is for assessment of chorea, dystonia, ataxia, extraocular movements, speech, gait, postural imbalance. Each subsection can be scored from 0-4. By summing up, the total score ranges from minimum 0 and maximum 124. Higher score means more severity.
Changes in spatiotemporal gait measures using objective gait analysis | 3 months
  The investigators will use Zeno Walkway Gait carpet and the spatiotemporal details of the gait will be analyzed by ProtoKinetics Movement Analysis Software (PKMAS) software, pre and post stimulation.The Zeno walkway will be used in conjunction with the ProtoKinetics Movement Analysis Software (PKMAS). The walkway contains a series of pressure sensors to detect footfalls. These data will be captured and collated via the PKMAS software, resulting in numerous spatial, temporal and pressure-related gait parameters. Timed-up-and-go (TUG) task will be used, consisting of rising from chair, walking across the 20-foot gait carpet, turning around off the carpet, walking back and sitting down.
Change in upper limb movements | 3 months
  The investigators will use KinArm pre and post stimulation to have objective measurement of upper limb movements. KinArm is a robotic manipulator arm. The patients will hold the manipulator arm and move it across to certain points shown on the computer screen. The investigators will use standard KinArm testing protocols to assess upper limb movements.
Change in speech | 3 months
  The investigators will use standardized speech protocol pre and post stimulation to assess speech. Participant's speech will be recorded using a head-mounted microphone (AKG-c520) and a digital recording device (Zoom H4nPro) while performing the following calibrated tasks. Calibration involves a sound level meter placed at 15cm from the mouth while talker says 'ah' at 70dBA. The following speech tasks will be assessed- Prolonged phonation, Rapid repetitions of the sounds, Two productions of a sentence with selected speech sounds, Two times louder production of a sentence with selected speech sounds, Repetition of a continuous vowel at normal and fast rates without making any voice breaks or pauses.
  f) Read aloud a section of a standard passage - standard rainbow passage g) Monologue. Talk for two minutes about an interesting vacation (or an interesting hobby or activity).
Changes in Network fragmentation using Quantitative EEG | 3 months
  The investigators will do network fragmentation by 5 mins of resting quantitative Electroencephalography (EEG), pre and post stimulation.Quantitative EEG signals will be recorded using g. Nautilus g.tec wireless system. The g. tech system uses ear clip reference sensors. Patient will sit in a comfortable arm chair in a quiet place with less light or electromagnetic perturbations. The patient will be instructed to sit relaxed with eyes closed for 5 min.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar S Jog, Principal Investigator — London Health Sciences Centre

REFERENCES:
- [Background] Eddy CM, Shapiro K, Clouter A, Hansen PC, Rickards HE. Transcranial direct current stimulation can enhance working memory in Huntington's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Jul 3;77:75-82. doi: 10.1016/j.pnpbp.2017.04.002. Epub 2017 Apr 5. PMID 28390970
- [Background] Berardelli A, Suppa A. Noninvasive brain stimulation in Huntington's disease. Handb Clin Neurol. 2013;116:555-60. doi: 10.1016/B978-0-444-53497-2.00044-9. PMID 24112923